CLINICAL TRIAL: NCT05641467
Title: The Effect Of Watchıng Vıdeo Wıth Vırtual Realıty Glasses On Paın, Anxıety And Satısfactıon Durıng Epızıotomy Repaır
Brief Title: Effect of Virtual Reality Glasses Use During Episiotomy Repair Related
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Rüveyde CAN, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0000-0002-1344-0908
Record Dates: First submitted 2022-11-09; First posted 2022-12-07 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Midwifery; Labor Delivery
Keywords: episiotomy; Virtual Reality; pain; satisfaction; anxiety
MeSH Terms: conditions — Pain; Personal Satisfaction; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Sample size G-power 3.1.9.7. program (Faul et al 2007, Faul et al 2009). Shourab et al. anxiety score average in the study; It was found to be 24.9±1.9 in the intervention group and 21.2±1.1 in the control group. In the light of this study, 0.897 effect size, 0.95 power, 0.05 alpha level and bidirectional hypothesis options were selected in the program, and the number of participants for each group was 34 (Shourab et al 2016). The pregnant women who came to the hospital will evaluate in terms of sample criteria and randomized sampling will divide into two groups. In order to ensure randomization in the study, a random numbers table was created by dividing them into two groups over the number determined on the site https://www.random.org/. Pregnant women will be assigned to groups according to the randomization scheme. Considering that there may be data loss, 20% more was determined and it was planned to study with 82 (41 intervention, 41 control) pregnant women.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video will be watched with virtual reality glasses during episiotomy repair (Experimental): Views of nature with virtual reality glasses during episiotomy repair.
  Interventions: Other: virtual reality glasses
- Control (No Intervention): It will be perform routine practice who the women in the control group.

INTERVENTIONS:
Other: virtual reality glasses — OculusQuest 2 128GB brand virtual reality glasses will be used in our research. OculusQuest 2 128GB is the original all-in-one gaming system for virtual reality. It can only be used as desired with the VR headset and controllers. It adapts to its environment. In this way, it can be played standing and sitting in small and large areas. When glasses will be used on another pregnant women within the scope of COVID-19 measures, disinfection will be provided with 'DiverseyOxivir Plus (hydrogen peroxide)' surface disinfectant. Before the episiotomy repair, the video glasses will be opened, the video will be adjusted to suit the woman. In order for the repair method to be the same for all women, It will be planned to use absorbable, synthetic, braided, sterile surgical thread produced from 1-0 polyglactin.
  Other Names: Video will be watched with virtual reality glasses during episiotomy repair
  Arms: Video will be watched with virtual reality glasses during episiotomy repair

SUMMARY:
H1-1: Watching video with virtual reality glasses during episiotomy repair reduces the level of pain.

H1-2 Watching video with virtual reality glasses during episiotomy repair reduces the level of anxiety.

H1-3: Watching video with virtual reality glasses during episiotomy repair increases the level of satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,

  * Able to speak Turkish and express himself in Turkish,
  * There is no visual or hearing impairment,
  * Being open to communication, spiritually and mentally healthy,
  * 37- 42 weeks of gestation
  * Single pregnancy,
  * Primiparity,
  * Vaginal delivery,
  * Vertexpresentation
  * Media lateral episiotomy,
  * Uncomplicated newborn
  * Newborns between 2500 and 4000 g.
  * Those with episiotomy between 4-8 cm

Exclusion Criteria:

* Presence of obstetric or non-obstetric complications,
* Presence of bleeding requiring urgent measures,
* Administration of sedative drugs before and during episiotomy repair, spinal anesthesia, epidural anesthesia, pudendal block (except for local infiltration of the perineum),
* Lacerations other than episiotomy (anal sphincter injury or Grade 3 or 4 tear),
* Instrument delivery (with vacuum or forceps),
* Postpartum complications in newborns,
* Chronic disease (diabetes mellitus, thyroid disease and hypertension),
* Having a psychiatric diagnosis

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 82 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
Socio-Demographic Data Collection Form | in active phase on labor (4 cm vaginal dilatation)
  Pregnant Introductory Information Form is a questionnaire prepared by researchers using the literature.
State-Trait Anxiety Inventory (STAI)-Questionnaire | immediately before repair episiotomy
  State-Trait Anxiety Inventory (STAI)-Questionnaire [ Time Frame: up to one hour ] STAI was used to measure the anxiety level of pregnant women. It was developed by Spielberger et al. (Spielberger et al., 1970) and Öner and Le Compte conducted a Turkish validity and reliability study of the scale (Öner & LeCompte, 1983). In the scale, individuals are provided to express their feelings with 40 expressions. With the state anxiety scale, it is possible to determine how the individual feels at the moment and in the conditions, and with the trait anxiety scale, how he feels outside of the current situation and conditions. The scale is a 4-point Likert type.The last score obtained shows the anxiety level of the individual. High scores from the scale indicate an increased level of anxiety, low scores indicate a decrease.
Visual Analog Scale-Pain (VAS-P) | immediately before repair episiotomy
  The VAS-P, which is used to evaluate the severity of pain, is a 10 cm long horizontally or vertically drawn ruler, starting with "No pain (0)" and ending with "Unbearable pain (10)". The woman is asked to show the point on this line that corresponds to the intensity of pain she feels. The distance between the marked point and the starting end of the line (0=no pain) is measured in centimeters and the numerical value found shows the severity of the patient's pain (Hayes and Patterson 1921). VAS-P is accepted as a safe, valid and usable measurement tool in repeated measurements. In this study, horizontally prepared VAS-P was used to assess pain intensity.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI)-Questionnaire | immediately after episiotomy repair
  State-Trait Anxiety Inventory (STAI)-Questionnaire [ Time Frame: up to one hour ]
Visual Analog Scale-Pain (VAS-P) | immediately after episiotomy repair
  The VAS-P, which is used to evaluate the severity of pain, is a 10 cm long horizontally or vertically drawn ruler, starting with "No pain (0)" and ending with "Unbearable pain (10)". The woman is asked to show the point on this line that corresponds to the intensity of pain she feels. The distance between the marked point and the starting end of the line (0=no pain) is measured in centimeters and the numerical value found shows the severity of the patient's pain (Hayes and Patterson 1921). VAS-P is accepted as a safe, valid and usable measurement tool in repeated measurements. In this study, horizontally prepared VAS-P was used to assess pain intensity.
Birth Action Follow-up Form | 60 minutes after birth
  This form includes the week of pregnancy, the height and weight of the pregnant woman, hemoglobin values, induction status, how long the birth stages last, the time of opening the episiotomy, the time of starting the repair, the ending time of the repair, the length of the episiotomy, the baby's Apgar score, the baby's weight.
Satisfaction Evaluation Scale and Form | immediately after episiotomy repair
  "Visual Analog Scale (VAS)" has been adapted to similar usage principles. The VAS is a scale that is evaluated by individuals on a horizontal or vertical line of 10 cm or 100 mm, with one end indicating that the individual is "very good" and the other end is "very bad".

CONTACTS AND LOCATIONS:
Overall Officials: Rüveyde Can, Principal Investigator — Necmettin Erbakan University, Faculty of Medicine
Locations (1):
- Fatma Deniz Sayıner, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No